CLINICAL TRIAL: NCT00703859
Title: A Phase I Single Arm Trial Combining Radiotherapy and Temozolomide With Dichloroacetate (DCA) in Patients With Newly Diagnosed Glioblastoma Multiform Tumours
Brief Title: Combining Radiotherapy and Temozolomide With Dichloroacetate in Patients With Newly Diagnosed Glioblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS-24139
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2011-09

CONDITIONS: Glioblastoma
Keywords: Radiotherapy plus temozolomide plus DCA; PK profile of DCA; MGMT promoter methylation status; Newly diagnosed Glioblastoma multiform tumours
MeSH Terms: conditions — Glioblastoma | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — DCA starting at an initial dose of 3mg/kg twice daily PO for consecutive days (days 1-5) on a 28 days cycle up to 6 cycles unless evidence of tumour progression. Each dose to be administered with food at the same time everyday 12 hours apart.

SUMMARY:
This is a study to see whether radiotherapy plus chemotherapy (Temozolomide) plus Dichloroacetate (DCA) improves overall survival and offers better control of the disease in patients with newly diagnosed Glioblastoma Multiforme Tumours.

DETAILED DESCRIPTION:
Patients with newly diagnosed Glioblastoma Multiforme Tumours, once consented to the study, would undergo standard treatment of radiotherapy plus chemotherapy (TMZ) with DCA in pill form (twice a day) during the radiation phase of the study and then with TMZ for six months after. Other elements of the clinical trial include pharmacokinetics and MGMT genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed GBM
* Diagnosis must be established by open biopsy or tumour resection
* Tumour must have a supratentorial component
* Over 18 years
* pre-treatment evaluations must be met
* study therapy to begin within 6 weeks of surgery
* KPS greater or equal to 70
* patients must sign informed consent
* If female, patients must not be pregnant or lactating
* Women of childbearing potential and male participants must practice adequate contraception

Exclusion Criteria:

* prior invasive malignancy )except for non-melanomatous skin cancer) unless disease free for greater than 3 years
* recurrent or multifocal malignant gliomas
* metastatic disease of leptomeningeal spread
* prior chemo or radiosensitizers for cancers of the head and neck region
* prior RT to head and neck region except for T1 glottic cancer, resulting in overlap of radiation fields.
* Severe active co-morbidity define in protocol
* Pregnant of lactating women
* Women of childbearing potential or men who are sexually active who are not willing or able to use medically acceptable forms of contraception; this exclusion is necessary due to the treatment involved potentially being teratogenic.
* prior allergic reaction to temozolomide and/or dichloroacetate
* History of HIV/AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of DCA in combination with radiotherapy and temozolomide in an adjuvant setting for the treatment of newly diagnosed GBM patients. | 2 years

SECONDARY OUTCOMES:
To determine if there is a correlation between MGMT promoter methylation status and progression-free survival for newly diagnosed GBM patients undergoing concurrent TMZ, DCA and RT followed by six monthly cycles of TMZ and DCA | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Abdulkarim, MD, FRCPC, Principal Investigator — AHS Cancer Control Alberta